CLINICAL TRIAL: NCT07344259
Title: Digital Health Literacy of Egyptian Parents and Its Association With Oral Health Outcomes of Their Preschool Children: An Analytical Cross-Sectional Study
Brief Title: Digital Health Literacy of Egyptian Parents and Oral Health Outcomes of Their Preschool Children
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatollah Nagy Sharkawy Ali Nada, Principal Investigator, Cairo University
Other Study IDs: CU 8.1.2026
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Digital Health Literacy; Caries Experience

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to examine the association between the digital health literacy (DHL) of Egyptian parents and oral health outcomes of their preschool children. The study will also examine the association between the parents' DHL and parents' sociodemographic characteristics. The main research question is:

What is the association between digital health literacy (DHL) of Egyptian parents and oral health outcomes of their preschool children?

DETAILED DESCRIPTION:
The study is an analytical cross-sectional study. It will involve Egyptian parents of preschool children to examine the association between their digital health literacy (DHL) and oral health outcomes of their preschool children. In addition, the study will assess the relationship between parents' DHL and sociodemographic characteristics.

Data will be collected using a structured questionnaire administered through face-to-face interviews or self-completed forms. The dimensions of digital health Literacy of the participants will be captured using the eHealth Literacy Questionnaire (eHLQ).

dmft scores will be recorded after clinical examination by trained dental health professionals.

Additionally, the questionnaire will include questions about sociodemographic data of parents and children, as well as dental habits of their children. All data will be coded, anonymized, and saved into a secure online database.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian parents or primary caregivers of at least one preschool aged child aged 3-5 years
* Willing to provide a consent for themselves and their child to participate in the study.

Exclusion Criteria:

* Individuals with cognitive impairments that limit their ability to complete the questionnaire.
* Individuals whose children have special care needs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Egyptian parents of preschool children attending a university hospital in Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Digital Health Literacy measured by E-Health Literacy questionnaire | The study will capture data at a single point from April -December 2026